CLINICAL TRIAL: NCT07001878
Title: Cannabis Potency Effects on Brain White Matter in Early Phase Psychosis: A Pilot Feasibility Treatment Study
Brief Title: Cannabis Potency Effects on Brain White Matter in Early Phase Psychosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Phil Tibbo, Principal Investigator, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 73219
Record Dates: First submitted 2025-05-07; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Psychosis; Cannabis Use
Keywords: cannabis; metformin; early phase psychosis; potency
MeSH Terms: conditions — Psychotic Disorders; Marijuana Abuse | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): All participants will receive 6 months of daily Metformin treatment and attend baseline, 3 months, and 6 months post baseline appointments.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be prescribed, reaching 1000mg/day (a standard dose). This will be done under the principal investigator's care and the patient's clinical team, including assessment of metformin adherence. Metformin will be prescribed for 6 months. Antipsychotic treatment will continue as per standard of care (metformin as adjunct therapy), as well as routine follow up.
  Other Names: Glucophage; Metformin Hydrochloride

SUMMARY:
Canada reports some of the highest rates of cannabis use in our youth and young adult populations, among all the developed countries. Recent Health Canada surveys report that 27% of 16-19-year-olds and 32% of 20-24-year-olds have used cannabis in the past 30 days, with 16-24-year-olds showing the highest rates of daily or near-daily use. Unfortunately, cannabis use has also been found to be a risk factor for the development of a psychotic disorder in emerging adults, and in those who develop psychosis and continue cannabis use, there is a significant effect on long term outcomes. This includes the severity of symptoms, risks of relapse (being hospitalized) and not reaching a level of functioning that would be expected. Lifetime experience with cannabis is greater than 80% in young adults with early phase psychosis (EPP; the first 5 years of a psychosis illness) with up to 30% of Canadian EPP patients meeting criteria for a diagnosis of cannabis use disorder (CUD) at entry to care. A recent Canadian population-based study found that cannabis use disorder associated to psychosis has risen from 3.7% pre-2018 to 10.3% at present. There has been a significant increase in Δ9-tetrahydrocannabinol (THC) levels in cannabis products available globally over the years, with popular cannabis products available start as high as 18% THC in Canada. However high potency cannabis carries a more significant risk for psychosis development, as well as higher risk for cannabis dependence and other severe mental health issues.

A major gap in the research is a specific focus on cannabis potency on brain white matter (WM) in youth and young adults, and if there are any potential treatment strategies that could be used to influence any of these cannabis WM effects. To address this, a medication called metformin, that is already used in psychosis to help with side effects of antipsychotic medications, will be used as it has also shown promise to influence WM changes in other illnesses. This project is thus focused on naturalistic cannabis potency effects on WM in emerging adults in EPP (divided into three groups; those using high potency cannabis, low potency cannabis, and minimal cannabis use) and treating them with metformin for 6 months and assessing effects on neuroimaging, cognitive and clinical variables.

The purpose of this pilot feasibility study is to inform the development/refinement of an intervention protocol, and not to test potential effects or mechanisms as the sample size will have insufficient power to perform an in-depth analysis. The results of this work will inform our research strategy development and assess feasibility of our novel methodological approach.

Participants will:

1. Visit the clinic at baseline, 3 months (only Timeline Follow-Back Assessment administered), and 6 months post baseline to complete substance use and mental health questionnaires, and cognitive assessments
2. Complete an MRI scan at baseline and 6 months
3. Take Metformin every day for 6 months

DETAILED DESCRIPTION:
Researchers will compare three groups of young adults with EPP: those using cannabis on a regular basis i) high potency (>15% THC) and ii) low potency (<15% THC) cannabis products and iii) patients with minimal-to-no cannabis use to see if there are differences in cannabis potency effects on white matter.

This study will collect four different types of variables: demographic (things that describe the participants), clinical (things that describe how ill the individuals are), substance use (things that measure how much or how reliant participants are on recreational substances), and neuropsychological (things that measure cognitive functioning such as attention, memory, verbal learning, and executive functioning).

Baseline demographics will include age, sex, gender and ethnicity. The Timeline Followback (TLFB) method will be used to collect detailed information about current cannabis use, which includes quantity, frequency, and potency (e.g., THC %, THC/CBD). Potency data will be self-report, verified whenever possible through the use of the Nova Scotia Liquor Corporation product website and other websites used for product purchase. Cannabis quantity and frequency will be assisted by visual aids. The TLFB has been validated for use among those with schizophrenia-spectrum disorders. The World Health Organization - Alcohol, Smoking, and Substance Involvement Screening Test (WHO-ASSIST) will be used to collect non-cannabis substance use data and the Cannabis Use Disorder Identification Test - Revised (CUDIT-R) will be used to measure problematic cannabis use. Overall psychosis symptoms will be measured by the Clinical Global Impression scale, for both severity and improvement (CGI-S, CGI-I). Cognitive data will be collected, focusing on tasks that are known to be affected by cannabis use (including high potency product). These include verbal learning and memory (California Verbal Learning Test-3; CVLT-3) and executive functioning (Trail Making Test B; TMT-B). In addition, the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) will be used which includes domains of immediate memory, language, attention, and delayed memory.

Neuroimaging: Subjects will undergo a Magnetic Resonance Imaging (MRI) scan collecting T1-weighted structural, diffusion-weighted scans and magnetic resonance spectroscopy data at baseline and 6 months post baseline.

Interim and final assessments: The TLFB will be completed 3 months post baseline. At 6-months post baseline, all the above measures and imaging will be repeated (study end).

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll individuals 18-25 years of age from the Nova Scotia Early Psychosis Program

Exclusion Criteria:

* Current stimulant use disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in cannabis use | Baseline, 3 months, 6 months
  Cannabis Timeline Followback (TLFB) is a retrospective past 30 day calendar method used to collect detailed information about current cannabis use, which includes quantity, method of use (e.g. dried cannabis smoked, concentrate vaped, edibles, etc.), frequency, strain, and potency (e.g., THC %, THC/CBD).
Treatment adherence | Baseline to 6 months
  The difference between the number of participants who completed 6 months of Metformin treatment compared to those who ceased using medication prior to study end at 6 months.
Change in white matter microstructure | Baseline to 6 Months
  Changes from baseline to study end at 6 months in study completers using Orientation dispersion index values from Neurite orientation dispersion and density imaging (NODDI).
Change in glial cell marker | Baseline to 6 months
  Measurement of glial cell marker neurochemical in the dorsomedial prefrontal region of brain Myo-inositol level changes from baseline to study end at 6 months for study completers using Magnetic resonance spectroscopy (MRS).
Recruitment success | Baseline
  The difference between the number of patients approached about the opportunity to participate and the total number of participants enrolled in the study for each study cohort.

SECONDARY OUTCOMES:
Change in white matter to grey matter ratio | Baseline to 6 months
  Changes from baseline in percent whole brain gray and white matter at 6 months assessed with MPRAGE imaging.
Change in inflammatory neurochemicals | Baseline to 6 months
  Measurement of inflammatory neurochemical changes in the dorsomedial prefrontal region of brain by measurement of total choline level changes in dorsomedial prefrontal region of the brain from baseline to 6 months using Magnetic resonance spectroscopy (MRS).
Change in overall substance use | Baseline to 6 months
  The WHO Alcohol, Smoking, and Substance Involvement Screening Test (WHO-ASSIST) will measure substance use risk scores to account for problematic use other than cannabis use from baseline to 6 months. Scores range from 0-39 for each substance with higher scores indicating more severe risk associated with use.
Changes in problematic cannabis use | Baseline to 6 months
  Cannabis Use Disorder Identification Test - Revised (CUDIT-R) will be used to measure problematic cannabis use scores from baseline to 6 months on a scale of 0-32 with higher scores indicating more problematic use.
Change in severity of illness | Baseline to 6 months
  Clinical Global Impression Scale - Severity (CGI-S) at baseline and then the complementary scale for follow-up the Clinical Global Impression Scale - Improvement (CGI-I) will measure changes from baseline in participants overall illness severity at 6 months, The CGI-S, a 7-point clinician rated Likert scale that measures individuals' overall illness severity relative those who the clinician has experienced with the same diagnosis (ranging from 1 = Normal, not at all ill to 7 = Extremely ill). The CGI-I is based on the CGI-S rating and is a 7-point clinician rated Likert scale ranging from 1 = Very much improved to 7 = Very much worse.
Changes in verbal learning | Baseline to 6 months
  The California Verbal Learning Test - Third Edition (CVLT3) will be used to measure changes in verbal learning index scores from baseline to 6 months. The CVLT3 measures episodic verbal learning including verbal learning, immediate memory, and delayed memory. The CVLT3 yields three index scores of overall verbal learning and memory performance using a mean of 100 and a standard deviation (SD) of 15 points. The scores range from 40-160, which is 4 SDs below and above the mean.
Changes in executive functioning | Baseline to 6 months
  Trail Making Test B (TMT-B) will be used to measure changes in recorded time taken to complete the task from baseline to 6 months. The assessment requires participant to draw a continuous line between circles containing letters and numbers in the correct ascending sequence (i.e., 1-A-2-B-3-C, etc.). Recorded test time more than 180 seconds indicates deficits in executive functioning.
Changes in overall cognitive functioning | Baseline to 6 months
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) will be used to measure changes in global cognition from baseline to 6 months. The RBANS is a comprehensive neuropsychological battery for the evaluation of global cognition and has been validated in subjects with schizophrenia. It includes measures of immediate and delayed memory, attention, visuospatial construction, and language. Scores range from 0 to 160 with 100 representing the population average. Higher scores represent better cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Tibbo, MD, Principal Investigator — Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and privacy considerations outlined by the Nova Scotia Health Authority. Data sharing was not a requirement of the study's funding, and given the small sample size, there is a heightened risk of re-identification of participants. To protect participant confidentiality and adhere to institutional ethics guidelines, data will remain securely stored and will not be made available to external parties.